CLINICAL TRIAL: NCT05558202
Title: Turkish Version of The Lower Limb Assessment Score : Reliability and Validity
Brief Title: Turkish Version of The Lower Limb Assessment Score
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emrah Afsar, Head of Occupational Therapy Deparment, Kutahya Health Sciences University
Other Study IDs: LLAS Study
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Hypermobility, Joint
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Turkish validity and reliability — 1. Explanation of the Turkish version of the scale.
  2. Translating the Turkish version of the scale into English to ensure consistency with the original scale.
  3. First application of scales to participants by two examiners separately.
  4. Second application of the scales to the participants by one examiner.
  5. Statistical analysis and scaling

SUMMARY:
Hypermobility is more than normal joint laxity, mobility, and range of motion. It is characterized by increased laxity and fragility of connective tissues. Symptoms from hypermobility can begin at any age and affect women more than men. People are at higher risk than other people. It is stated that hypermobility is an important factor in orthopedic injuries and diseases. Individuals with hypermobility have more frequent orthopedic complaints and the problems are usually idiopathic and chronic. Studies have reported that proprioception and musculoskeletal reflex function may be affected independently of symptoms in hypermobile individuals. Therefore, evaluating hypermobility is very important in preventing hypermobility-related problems and injuries and developing appropriate treatment methods. Although the Beighton score is the most commonly used scoring method to determine hypermobility, it may be insufficient to determine hypermobility of the lower extremities. The Lower Limb Assessment Score (LLAS) has been reported to be one of the most appropriate scoring methods for assessing lower extremity hypermobility in the literature. The aim of this study is to adapt LLAS to Turkish and measure its validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged between 18 to 35

Exclusion Criteria:

* Using assistive devices or orthoses for the upper extremity
* Surgery history of the upper extremity
* Pain located on the upper extremity in the last 6 months
* Previous trauma that might restrict normal range of motion.
* Having degenerative or inflamatuar disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: - The study will be carried out by young adults and adults in the Kutahya Health Science University
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The Lower Limb Assessment Score (LLAS) | 10 minutes
  The LLAS was designed to test the mobility of many joints of the lower limb in multiple planes of motion. These tests include passive physiological, passive accessory and active range of motion.
  The LLAS is performed on both lower limbs, each providing a score to a maximum of 12.
The Beighton Score | 5 minutes
  The Beighton Score is a set of manoeuvres used as the standard method of assessment for Generalised Joint Hypermobility. The Beighton score arbitrarily investigates the presence of hyperlaxity (yes = 1, no = 0) at both wrists, the fifth metacarpo-phalangeal joints, elbows, knee joints, and the lumbosacral spine. The items are summed and yield a Beighton score ranging from 0 to 9 points.

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Afsar, Phd, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No